CLINICAL TRIAL: NCT04477343
Title: An Open-label Phase 1 Study to Evaluate the Safety and Tolerability of SX-682 in Combination With Nivolumab as a Maintenance Therapy in Patients With Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: A Study to Evaluate the Safety and Tolerability of SX-682 in Combination With Nivolumab as a Maintenance Therapy in Patients With Metastatic Pancreatic Ductal Adenocarcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Syntrix Biosystems, Inc. (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Daniel Mulkerin, Professor - Department of Medicine , Hematology/Oncology, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UGIP20027
Record Dates: First submitted 2020-07-10; First posted 2020-07-20 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer
Keywords: Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental: SX-682 and Nivolumab (Experimental): SX-682 Dose: 25, 50, 100, 200, 400mg BID taken as an oral pill
  Nivolumab Dose: 240mg, every 2 weeks via intravenous infusion
  Interventions: Drug: SX-682; Drug: Nivolumab Injectable Product

INTERVENTIONS:
Drug: SX-682 — Allosteric inhibitor to human CXCR1 and CXCR2 receptor
Drug: Nivolumab Injectable Product — humanized monoclonal antibody to program cell death receptor 1 (PD1)

SUMMARY:
The main purpose of this research study is to determine the maximum tolerable dose (MTD) of SX-682 in combination with nivolumab in patients with metastatic pancreatic ductal adenocarcinoma who have completed at least 16 weeks of first line chemotherapy treatment without evidence of disease progression.

DETAILED DESCRIPTION:
In this study the investigator would like to better understand the maximum tolerable dose (MTD) of SX-682 in combination with nivolumab in patients with metastatic pancreatic ductal adenocarcinoma who have completed at least 16 weeks of first line chemotherapy treatment without evidence of disease progression. In addition, the investigator would like to measure the SX-682 pharmacokinetic data in humans. The investigator would also like to assess the immunophenotypic and stromal changes to the tumor microenvironment after treatment.

ELIGIBILITY:
Inclusion Criteria:

Written Informed Consent and HIPAA Authorization

1. Subjects must have the nature of the study explained to them
2. Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, pharmacokinetic collections, study biopsies and other requirements of the study.
3. Subjects (or an acceptable proxy) must provide a signed and dated IRB/IEC approved written informed consent form (ICF) in accordance with regulatory and institutional guidelines for both the study and exploratory biomarker analysis obtained via paired biopsies.
4. Subjects (or an acceptable proxy) must provide a signed and dated Health Insurance Portability and Accountability Act (HIPAA) authorization.
5. The ICF and HIPAA authorization must be obtained before conduction and procedures that do not form a part of the subject's normal care.
6. After signing the ICF and HIPAA Authorization, subjects will be evaluated for study eligibility during the Screening Period (no more than 28 days before study drug administration) according to the following further inclusion/exclusion criteria:

Study Population/Inclusion Criteria

1. Male or female subjects, aged at least 18 years
2. Have histologically or cytologically confirmed metastatic pancreatic ductal adenocarcinoma
3. Completion of at least 16 weeks of first line chemotherapy without evidence of disease progression
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
5. Must have measurable disease with at least 1 unidimensional measurable lesion per iRECIST
6. Screening laboratory values within 14 days prior to first dose of study drug:

   WBC ≥ 3000/µL Neutrophils ≥ 1500/µL Platelets ≥ 100,000>µL Hemoglobin ≥ 9.0 g/dL in the absence of blood transfusion Creatinine ≤ 1.5 mg/dL AST/ALT ≤ 2.5 x ULN for subjects with no liver metastases
   * 5 x ULN for subjects with liver metastases Bilirubin ≤ 1.5 mg/dL sa≤ 3.0 mg/dL for subjects with Gilbert's disease INR or PT ≤ 1.5 x ULN unless receiving anticoagulation therapy aPTT or PTT ≤ 1.5 x ULN unless receiving anticoagulation therapy
7. Life expectancy of ≥ 12 weeks as judged by the treating physician.
8. Patient must consent for baseline and on treatment biopsies
9. Patients must have baseline pulse oximetry ≥ 90% on room air

Exclusion Criteria:

Target Disease Exceptions:

Active brain metastases or leptomeningeal metastases. Subjects with brain metastases are eligible if these have been treated and there is no magnetic resonance imaging (MRI- except where contraindicated, in which case a CT scan is acceptable) evidence of progression for at least 8 weeks after treatment is complete and within 28 days prior to first dose of study drug administration. An MRI is not required to rule out brain metastases or leptomeningeal metastases. There must also be no requirement for high doses of systemic corticosteroids that could result in immunosuppression (>10 mg/day prednisone equivalents) for at least 2 weeks prior to study dry administration.

Medical History and Concurrent Disease

Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results. Specifically:

1. Subjects with active, non-infectious pneumonitis.
2. Subjects with interstitial lung disease or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management.
3. Subjects with clinically significant heart disease that affects normal activities.
4. Clinically significant cardiovascular/ cerebrovascular disease defined as cerebral vascular accident, stroke, carotid artery disease transient ischemic attach (< 6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association Classification Class >II) or serious cardiac arrhythmia.
5. Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix or breast.
6. Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
7. Subjects with a condition (including organ or bone marrow transplant) requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
8. Use of other investigational drugs (drugs not marketed for any indication) or medications at immunosuppressive doses within 28 days before study drug administration.
9. Patients who received immunotherapy or investigational drug within 4 weeks prior to enrollment.
10. Patients who underwent major surgery within 4 weeks of enrollment (not including diagnostic laparoscopy)
11. History of myelodysplastic syndromes or myeloproliferative neoplasms.
12. History of or medication induced prolonged QT interval.
13. Any botanical preparation (e.g., herbal supplements or traditional Chinese medicines) intended to treat the disease under study or provide supportive care. Use of marijuana and its derivatives for treatment of symptoms related to cancer treatment, even if obtained by medical prescription or if its use (even without a medical prescription) has been legalized locally.

Physical and Laboratory Test Findings

1. A history of Hepatitis B or C, either acute or chronic, as indicated by HBV surface antigen positivity, HBV core antibody positivity, or positive HCV antibody with reflex to positive HCV RNA.
2. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
3. Active tuberculosis (history of exposure or history of positive tuberculosis test plus presence of clinical symptoms, physical or radiographic findings).
4. EKG demonstrating a QTc interval >470 msec or patients with congenital long QT syndrome.

Allergies and Adverse Drug Reaction

1. History of allergy to study drug components (examples: hydroxpropylmethylcellulose phthalate (hypromellose phthalate or HPMCP), microcrystalline cellulose, sodium croscarmellose, sodium lauryl sulfate, and silicon dioxide).
2. History of severe hypersensitivity reaction to any monoclonal antibody (Grade ≥ 3 NCI-CTCAE v5).
3. History of anaphylaxis, or recent (within 5 months) history of uncontrolled asthma.

Sex and Reproductive Status/Special Populations

1. Women of childbearing potential (WOCBP) must use method(s) of contraception with a failure rate of less than 1% while on study and for 5 months after the last dose of SX-682 or nivolumab. A WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over age 45 in the absence of other biological or physiological causes.
2. Women under the age of 62 with a history of being postmenopausal must have a documented serum follicle stimulating hormone, (FSH) level > 40 mIU/mL.
3. Women must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug.
4. Women must not be breastfeeding.
5. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year while on study and for a period at least 7 months after the last dose of study drug.
6. Women who are not of childbearing potential and azoospermic men do not require contraception.
7. Individuals who are incarcerated, compulsory detained or otherwise considered a vulnerable population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-11-23 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerable dose [Safety and Tolerability] | through study completion, an average of 6 months
  Maximum tolerable dose is defined by less than or equal to 30% dose limiting toxicity (DLT) event rate within a given dose combination,

SECONDARY OUTCOMES:
Progression Free Survival | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Measure of time from study enrollment until progression.
Overall Survival | From date of enrollment until date of death from any cause up to 24 months
  Measure of time from study enrollment until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Mulkerin, MD, Principal Investigator — University of Rochester Wilmot Cancer Center
Locations (1):
- University of Rochester, Rochester, New York, United States